CLINICAL TRIAL: NCT00423774
Title: A Feasibility Study to Test an Individualized Dyadic Problem-Solving Education Intervention to Improve Problem-Solving Skills of Patients and Family Caregivers During Allogeneic HSCT
Brief Title: Education Program to Manage Emotional Stress of Stem Cell Transplant Recipients and Their Caregivers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 070067; 07-CC-0067
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-28

CONDITIONS: Family Caregivers; Bone Marrow Transplantation
Keywords: Allogeneic Hematopoietic Stem Cell Transplant; Psychological Distress; Coping; Cognitive Behavior Therapy; Bone Marrow Transplant; Coping Skills

INTERVENTIONS:
Behavioral: Problem-Solving Education

SUMMARY:
his study will evaluate a series of problem-solving education sessions for patients undergoing a stem cell transplant and their family caregivers. The emotional stress of transplant extends beyond patients to their families, especially caregivers. Little is known about managing the emotional distress associated with stem cell transplant or the support and education most helpful to caregivers of stem cell recipients.

Patients undergoing a stem cell transplant and their family caregivers may be eligible for this study. All participants must be 18 years of age and older.

Patients and their caregivers receive routine treatment-specific education from transplant team members. This study adds a series of educational sessions focusing on problem-solving skills. In addition to the study education, participants do the following:

* Complete a 130-item questionnaire when they consent to participate in the study.
* Complete a 60-item questionnaire and attend a 60-minute face-to-face education session before the transplant.
* Complete a 40-item questionnaire and attend a 60-minute face-to-face education session before hospital discharge.
* Complete the same 40-item questionnaire and attend a 60-minute face-to-face education session 2 weeks after hospital discharge.
* Attend a 30-minute face-to-face education session 4 weeks after hospital discharge.
* Complete a 60-item questionnaire 6 weeks after hospital discharge.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HSCT) generates multiple symptoms and problems that can vary in complexity. Although it seems evident that patients and caregivers experience clinically significant levels of psychological distress, few intervention studies have been explored to address this concern in this population.

Problem-solving is an essential skill for patients and caregivers. Increased problem-solving skill has been shown to decrease psychological distress and may improve symptom distress and health related QOL. The COPE (Creativity, Optimism, Planning, Expert Information) problem-solving education intervention has demonstrated benefit and has been reported as a positive therapy by cancer patients and their families. Only one study has reported the application of this intervention in the acute care setting and no study has been done with patients undergoing allogeneic HSCT.

This study will evaluate the feasibility of conducting an individualized dyadic problem-solving education (PSE) intervention in patients and family caregivers experiencing allogeneic HSCT. In addition, this study will explore the effect of a PSE intervention on problem-solving skills in patients and family caregivers experiencing allogeneic HSCT. Moreover, this study will explore the relationship of baseline psychological distress and family functioning to change in problem-solving skills following a PSE intervention.

This is a single group, mixed-methods, repeated measure design. Subjects will be accrued to this protocol if they agree to participation in an allogeneic HSCT at the Clinical Center, NIH, are greater than or equal to 18 years old, able to read English and able to comprehend the investigational nature of the study. Patient volunteers must have an adult family member to serve as their primary caregiver throughout the study period. A sample of 20 subjects (10 patient/family caregiver dyads) will be recruited to capture the essence of the experience and adequately evaluate the feasibility of the intervention in this sample.

Each dyad will be scheduled for four individualized PSE intervention sessions (study intervention) in addition to the usual care group education. Study questionnaires will be administered twice prior to allogeneic HSCT, at 2 time points during the intervention period, and at the end of the study. As a feasibility study, there will be no long term follow-up after the intervention period. Questionnaires include: Brief Symptom Inventory-18, Problem-Solving Inventory-Revised, Symptom Distress Scale, and the Family Adaptability-Cohesion Evaluation Scale-IV. In addition, the dyad will participate in a semi-structured interview at the end of each intervention session and the interventionist will complete a log that tracks subject attendance, session length, and discrepancy between planned and actual session date and time. Quantitative and qualitative analysis techniques will be used in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients: Receiving their first allogeneic HSCT at the CC, NIH

Age greater than or equal to 18 years old.

Ability to comprehend the investigational nature of the study and provide informed consent.

Able to read and speak English.

Adult family member serves as primary caregiver throughout study period.*

Family caregiver agrees to participate in the study.

Family Caregiver (FC):

Age greater than or equal to 18 years old.

Ability to comprehend the investigational nature of the study and provide informed consent.

Able to read and speak English.

Adult family member who meets the patient inclusion criteria.

Family member (patient) agrees to participate in the study.

Intends to serve as primary caregiver throughout study period*

*If the FC changes during the study, the PSE intervention will continue as scheduled with the new FC, however, FC data will no longer be collected and will be excluded from the analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01-11; Primary Completion 2008-12-01 (Actual); Study Completion 2008-12-01 (Actual)

PRIMARY OUTCOMES:
Participation themes and implementation variances

SECONDARY OUTCOMES:
Problem solving skills in patient and caregiver

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldman JM, Horowitz MM. The international bone marrow transplant registry. Int J Hematol. 2002 Aug;76 Suppl 1:393-7. doi: 10.1007/BF03165291. PMID 12430889
- [Background] Thomas ED, Blume KG. Historical markers in the development of allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 1999;5(6):341-6. doi: 10.1016/s1083-8791(99)70010-8. No abstract available. PMID 10595811
- [Background] Tabbara IA, Zimmerman K, Morgan C, Nahleh Z. Allogeneic hematopoietic stem cell transplantation: complications and results. Arch Intern Med. 2002 Jul 22;162(14):1558-66. doi: 10.1001/archinte.162.14.1558. PMID 12123398